CLINICAL TRIAL: NCT03771586
Title: A Phase 1, Double-blind, Placebo-controlled Crossover Study of SAGE-718 Using a Ketamine Challenge, to Evaluate the Electrophysiology, Safety, Tolerability, and Pharmacokinetics in Healthy Subjects
Brief Title: A Study to Assess the Electrophysiology, Safety, Tolerability, and Pharmacokinetics of SAGE-718 Using a Ketamine Challenge in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 718-EXM-101
Record Dates: First submitted 2018-10-02; First posted 2018-12-11 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2022-01

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAGE-718 (Experimental)
  Interventions: Drug: SAGE-718
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAGE-718 — SAGE-718 in combination with Ketamine
  Other Names: Ketamine
  Arms: SAGE-718
Drug: Placebo — Placebo in combination with Ketamine
  Arms: Placebo

SUMMARY:
This study is a phase 1, double-blind, placebo-controlled crossover study of single, oral dose of SAGE-718 using a ketamine challenge, to evaluate the electrophysiology, safety, tolerability, and pharmacokinetics in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a body weight ≥50 kg and body mass index ≥18.0 and ≤30.0 kg/m2 at screening.
2. If female, subject is post-menopausal (at least 12 months of spontaneous amenorrhea with confirmatory follicle stimulating hormone >40 mIU/mL), or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, and/or hysterectomy).
3. Subject is healthy with no history or evidence of clinically relevant medical disorders as determined by the Investigator.

Exclusion Criteria:

1. Subject has a history or presence of any psychiatric disease or condition including suicidal ideation or behavior, has answered YES to any question on the C-SSRS at screening or admission, or is currently at risk of suicide in the opinion of the Investigator.
2. Subject has a history or presence of a neurologic disease or condition, including but not limited to epilepsy, closed head trauma with clinically significant sequelae, or a prior seizure.
3. Subject has a family history of epilepsy.
4. Subject has obstructed venous access and/or has skin disease, rash, acne, or abrasion at venous access site that may affect the ability to obtain a PK sample or affect the ability to receive the ketamine infusions.
5. Subject has had previous exposure to or is known to be allergic to ketamine or any of its excipients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2019-01-02 (Actual)

PRIMARY OUTCOMES:
Change in the electrophysiological parameters, auditory evoked potentials, between pre- and post-ketamine infusion in subjects receiving SAGE-718 vs the change in parameters between pre- and post-ketamine infusion in subjects receiving placebo | Between Day 1 and Day 11

SECONDARY OUTCOMES:
Safety and tolerability of SAGE-718-alone and in combination with ketamine, as assessed by the incidence of adverse events (AEs)/serious AEs (SAEs). | Between Baseline and Day 27
Safety and tolerability of SAGE-718-alone and in combination with ketamine, as assessed by changes from baseline in 12-lead electrocardiograms (ECGs) including PR interval, QT interval, QTc interval, QTcF, and rhythm abnormalities | Between Baseline and Day 12
  Observed values and change from baseline in ECGs in patients post study drug administration
Safety and tolerability of SAGE-718-alone and in combination with ketamine, as assessed by changes from baseline in electroencephalograms (EEGs) including Delta, Theta, Alpha, Beta. | Between Baseline and Day 12
  Observed values and change from baseline in EEGs in patients post study drug administration
Safety and tolerability of SAGE-718-alone and in combination with ketamine, as assessed by changes from baseline in Columbia-Suicide Severity Rating Scale (C-SSRS). | Between Baseline and 27 days
Safety and tolerability of SAGE-718-alone and in combination with ketamine, as assessed by changes from baseline in Brief Psychiatric Rating Scale (BPRS). | Between Day 1 and Day 11
Safety and tolerability of SAGE-718-alone and in combination with ketamine, as assessed by changes from baseline in Clinician Administered Dissociative State Scale (CADSS). | Between Day 1 and Day 11
Safety and tolerability of SAGE-718-alone and in combination with ketamine, as assessed by changes from baseline in Observer's Assessment of Alertness and Sedation (OAAS). | Between Day 1 and Day 11

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Sage Investigational Site, Long Beach, California
  - Sage Investigational Site, Berlin, New Jersey

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.

REFERENCES:
- See also: Related Info — http://www.sagerx.com